CLINICAL TRIAL: NCT02306434
Title: Fear of Childbirth - Comparison of Two Treatment Options: Internet Given Behavioral Therapy and Counseling by Midwife- a Clinical Randomized Controlled Trial
Brief Title: Fear of Childbirth - Comparison of Two Treatments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Mid Sweden University (Other); University of Melbourne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U-CARE: Pregnancy
Record Dates: First submitted 2014-12-01; First posted 2014-12-03 (Estimated); Last update posted 2018-04-13 (Actual); Status verified 2018-04

CONDITIONS: Fear of Childbirth; Pregnancy
Keywords: childbirth fear; Internet CBT; counselling; antenatal care; postnatal care; childbirth; Cognitive behavioural therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Therapy by iCBT (Active Comparator): Internet Cognitive behavioral therapy (iCBT) is given by a psychologist in the U-CARE platform. The intervention will focus on management of childbirth related fear. This means that the participants read texts and do homework assignments instructed from an internet page. Additional resources such as pictures, animations, videos and sounds will be a part of the treatment program. A psychologist will communicate with the participants through internal text-messages and will give feed back on their home work assignments. The content of the intervention will be standard components from CBT, for example relaxation training, behavioral activation, exposure for fear related stimuli, cognitive restructuring, behavioral sleep treatment.
  Interventions: Behavioral: Therapy by iCBT
- Standard care-Counselling (Other): Counselling for childbirth fear is given by the antenatal care midwife and by specially trained midwives working in collaboration with obstetricians at approximately 3-5 face to face counselling sessions. Often a visit to the delivery unit is included in the program and a care plan for the coming birth.
  Interventions: Other: Standard care-counselling

INTERVENTIONS:
Behavioral: Therapy by iCBT — Internet Cognitive behavioral therapy (iCBT) is given by a psychologist in the U-CARE platform. The intervention will focus on management of childbirth related fear. This means that the participants read texts and do homework assignments instructed from an internet page. Additional resources such as pictures, animations, videos and sounds will be a part of the treatment program. A psychologist will communicate with the participants through internal text-messages and will give feed back on their home work assignments. The content of the intervention will be standard components from CBT, for example relaxation training, behavioral activation, exposure for fear related stimuli, cognitive restructuring, behavioral sleep treatment.
  Other Names: Internet based Cognitive behavioural therapy
  Arms: Therapy by iCBT
Other: Standard care-counselling — Standard care (Counselling by midwives)
  Arms: Standard care-Counselling

SUMMARY:
Childbirth related fear is a public health issue strongly related to subsequent reproduction, a request for caesarean section and women's and children's health. Currently, women are offered 3-5 counseling sessions with specially trained midwives and obstetricians in most Swedish hospitals as standard care (SC). In general, women are satisfied with counseling but research show no major effect on cesarean section rates neither in decreased level of childbirth related fear. It is therefore important to find the best available treatment for this issue.

The aim of this program is to compare Internet given cognitive behavior therapy (ICBT) with standard counseling care for pregnant women reporting childbirth related fear.

Research questions: What effect does ICBT compared to SC have on a) the level of childbirth related fear b) a request for cesarean section c) compliance and satisfaction with treatment.

Design: A randomized controlled trial of women reporting childbirth related fear during pregnancy. One arm will receive SC and one arm ICBT though the U-CARE platform. Follow up of given treatment will occur at 30 and 36 weeks of pregnancy, two months and one year after birth. Intervention: The intervention will focus on management of childbirth related fear. This means that the participants do weekly sessions and homework assignments during pregnancy.

Primary outcome will be level of childbirth related fear measured at 36 weeks of pregnancy.

Secondary outcomes are level of childbirth related fear at 2 months and one year after birth, preferences for mode of birth, request for elective cesarean section, compliance and satisfaction with treatment and costs.

Expected benefits: This study will contribute to the development of new treatment methods for childbirth related fear. Evidence of the best treatment to reduce childbirth related fear based on the results from this study could be implemented in clinical practice and hopefully decreases the numbers of cesarean sections without medical indications.

DETAILED DESCRIPTION:
Project area

Childbirth related fear is a public health issue strongly related to subsequent reproduction and women's and children's health. It could be assumed that previous negative birth experiences are caused by interventions and/or lack of support from staff during birth which in turn could be linked to women's emotional wellbeing. Childbirth related fear often involves a request for a caesarean section, which in turn could have short and long term consequences for women's and children's health. The majority of studies on childbirth related fear have focused on maternal characteristics and the reasons for childbirth fear. Fewer studies have addressed treatment options for curing childbirth fear. Standard care for women with childbirth related fear in Sweden, is usually counseling with midwives and sometimes this counseling leads to an elective caesarean section. In general, women are satisfied with counselling. However, research shows no major effect of counselling, neither in decreased numbers of cesarean sections on maternal request nor in decreased levels of childbirth related fear one year after birth. Today a substantial financial amount of the budget for women's health care is allocated to treatment of childbirth fear using counselling teams. The introduction of such counseling teams was introduced without being preceded by any randomized trials about its effects. In other areas of health care, cognitive behavior therapy is recommended for psychosocial issues. The present project will compare Internet based cognitive behavior therapy (iCBT) with standard care (SC).

Survey of the field Childbirth related fear has gained major research interest particularly in the Scandinavian countries.Severe fear of childbirth has been reported to 6-10% in a Finish study, and fear comparable to PTSD 1.3%. Measures of childbirth related fear: The FOBS scale was developed in a cross-cultural comparative study where two VAS scales (measuring worries and fears in relation to childbirth) were combined.

Reported reasons for fear of childbirth are; fear of pain, childhood abuse, and feelings that the woman or the baby will be damaged during birth or even die, being denied help from caregivers or felt badly treated by delivery staff and, for multiparous women previous emergency caesarean sections or previous negative experiences of birth.

Treatment for childbirth fear Most Swedish hospitals have special counseling teams for women with childbirth fear, often called Aurora groups. Their antenatal midwife refers women to these special teams. The most common treatment model for these women are visits with a specially trained midwife, but psycho-somatic support, cognitive behavior therapy, and relaxation techniques are also used. This counseling treatment in Sweden has not been preceded by large randomized studies, but studies indicate that women are satisfied with the treatment. It has also been shown that women who are referred to the Aurora services more frequently have caesarean sections.

Aim and research questions The aim of this study is to compare Internet given cognitive behavior therapy (ICBT) with standard care (SC) for pregnant women identified with childbirth related fear.

Research questions: What effect does Internet given cognitive behavior therapy compare to standard care have on a) the level of childbirth related fear b) request for cesarean section c) compliance and satisfaction with care and d) costs for the treatment?

Method

Design: A randomized controlled trial of women with childbirth related fear. One arm will receive standard care and one arm cognitive behavioral therapy by internet.

Setting: One large Swedish university hospital and two regional hospitals. Recruitment: All pregnant women at the routine ultrasound screening examination, offered to all pregnant women during gestational week 16-20, will receive oral and written information about the study. The recruitment process will follow two steps. First, all women who attend the ultrasound examination will be handed a leaflet where a few questions are asked about their age, parity, gestational week, access to Internet and the FOBS-scale. The women will receive a brief information text with information about the purpose of the study, e.g. that we are interested in women's feelings towards the approaching birth and if they score over the cutoff point will be offered to attend a study of treatment for childbirth fear. To be eligible for inclusion, potential participants have to meet the following criteria; a) Swedish speaking b) scoring ≥60 on the FOBS score c) available internet access.

In the second step of recruitment, women who score 60 or above on the FOBS-scale will be sent a letter of invitation and a phone call from the recruiting midwives. The invitation letter and the phone call will explain the study outline and the women will be informed that they will be randomized either to iCBT or standard care. Informed consent from the women will be returned either by an on-line form to the U-CARE platform or in a prepaid envelope indicating consent or not. The women will be provided with login details to the U-CARE platform and all communication thereafter will be though the platform regardless of which arm women will be randomized to. After completion of a baseline questionnaire randomization to treatment will occur and women will receive instructions about the following program. If randomized to the iCBT arm the psychologist will introduce the iCBT-treatment by a telephone call.

Intervention: Internet Cognitive behavioral therapy (iCBT) is given by a psychologist by the U-CARE platform. The intervention will focus on management of childbirth related fear. This means that the participants read texts and do homework assignments instructed from an internet page. Additional resources such as pictures, animations, videos and sounds will be a part of the treatment program. A psychologist will communicate with the participants through internal text-messages and feed back on their homework assignments.The therapist will devote time to each participant each week via the Internet. The content of the intervention will be standard components from CBT, for example relaxation training, behavioral activation, exposure for fear related stimuli, cognitive restructuring, behavioral sleep treatment. The women complete homework assignments, this consists of tasks such as doing relaxation training, to perform planned new behaviors, to break behavioral habits, to expose oneself to frightening situations or to change sleeping routines.

Standard care: Counselling for childbirth fear is given by the antenatal care midwife and by specially trained midwives working in collaboration with obstetricians at approximately 3-5 face to face counselling sessions. Often a visit to the delivery unit is included in the program.

Measures: At baseline previously validated instruments measuring women's levels of fear of childbirth, anxiety, depressive symptoms, stressful life events, Prenatal Attachment Inventory (PAI-R), Blood and injection phobia, Cambridge Worry Scale, Performance Based Self-esteem, and Pain Catastrophizing scale.

In addition to the instruments included, women's socio-demographic and obstetrics background, psychosocial history, experience of childbirth, attitudes towards birth, partner and family support will be measured along with the woman's previous birth preferences.

Follow up: The randomized women will receive follow up questionnaires at 30 and 36 weeks of pregnancy where women's fears and emotional wellbeing will be further investigated using the above mentioned instruments. Two months and one year after birth additional questions about birth outcome, birth experience, breast feeding duration, attachment and bonding to their infant and their satisfaction and experience of the treatment program.

Outcome measures: The primary outcome will be level of childbirth related fear at 36 weeks gestation. Secondary outcomes are childbirth related fear at two months and one year after birth, preferences for mode of birth, request for cesarean section in late pregnancy and in case of a subsequent pregnancy, compliance and satisfaction with the treatment, birth outcome and costs.

Power analysis: A previous Swedish study showed that 59% of women with childbirth fear during pregnancy were 'cured' after a year. A power calculation based on a 20% reduction in childbirth fear, a two-sided test, a power of 0.80 and a level of significance of 5 %, shows that approximately 200 women need to be enrolled in the study.

Ethical considerations: The study has received full ethical review and approval. The hospital managers at the participating sites are cooperating with the study. The project leaders' name and contact details are available in the letter of invitation and women as well as recruiting midwives are encouraged to make contact if they have questions about the project. All data collection will be administered by the U-CARE platform and the research group.

Justification: Fear of childbirth is a public health issue strongly related to subsequent reproduction and women's and children's health. Currently identification and treatment is taking place without a clear evidence base. It is therefore important to find the most effective and acceptable treatment for this issue which can be offered to the maximum number of affected women in the most cost effective and sustainable manner. The study is linked to new innovations in person centered care in clinical practice using Internet based technology which is offering new and equitable access to best practice health care.

Expected benefits: This study will contribute to the development of new treatment methods for childbirth related fear. Finding evidence of the best treatment to reduce childbirth related fear based on the results from this study could be implemented in clinical practice and hopefully reduces the psychological distress felt by women during the childbearing period and reduces the number of caesarean sections requested by women without medical indications.

Consumer perspective and disseminating of study results: Prior to the recruitment of study participants think-aloud interviews with approximately 30 women will be performed in order to test the included instruments. In the pilot study women will carefully answer all questions and at the same time communicate their thoughts to a researcher when completing the questions, for construct and face validity.

ELIGIBILITY:
Inclusion Criteria:

* Mastery of the Swedish language,
* FOBS above 60,
* internet access

Exclusion Criteria:

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2014-03; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Level of childbirth related fear (FOBS) | 36 weeks of gestation
  Level of childbirth related fear

SECONDARY OUTCOMES:
Level of childbirth related fear (FOBS) | 2 months post-partum
  Level of childbirth related fear
Level of childbirth related fear (FOBS) | 1 year post-partum
  Level of childbirth related fear
Preferred mode of birth (vaginal or cesarean section) | 36 weeks of gestation
  vaginal or cesarean section
Request for cesarean section (yes or no) | 1 year postpartum
  yes or no

OTHER OUTCOMES:
Compliance with treatment (Number of treatments and satisfaction) | 2 month postpartum
  Number of treatments and satisfaction
Compliance with treatment (Number of treatments and satisfaction) | 1 year postpartum
  Number of treatments and satisfaction
Costs (SEK (Swedish currency) | 1 year postpartum
  SEK (Swedish currency)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Rubertsson, Ass Prof, Principal Investigator — Uppsala University Hospital
Locations (1):
- Uppsala university, Uppsala, Sweden

REFERENCES:
- [Derived] O'Connell MA, Khashan AS, Leahy-Warren P, Stewart F, O'Neill SM. Interventions for fear of childbirth including tocophobia. Cochrane Database Syst Rev. 2021 Jul 7;7(7):CD013321. doi: 10.1002/14651858.CD013321.pub2. PMID 34231203
- [Derived] Rondung E, Ternstrom E, Hildingsson I, Haines HM, Sundin O, Ekdahl J, Karlstrom A, Larsson B, Segeblad B, Baylis R, Rubertsson C. Comparing Internet-Based Cognitive Behavioral Therapy With Standard Care for Women With Fear of Birth: Randomized Controlled Trial. JMIR Ment Health. 2018 Aug 10;5(3):e10420. doi: 10.2196/10420. PMID 30097422
- See also: A randomized controlled study comparing internet-based cognitive — http://dx.doi.org/10.1016/j.srhc.2017.06.001